CLINICAL TRIAL: NCT01930877
Title: The Effect of Perioperative Lidocaine on Postoperative Quality of Recovery in Patients Undergoing Spine Surgery: A Randomized, Double - Blinded, Placebo Controlled Study
Brief Title: Effect of Perioperative Intravenous Lidocaine on Postoperative Quality of Recovery in Patients Undergoing Spine Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn by PI
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Suman Rajagopalan, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-32510
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Pain
Keywords: quality of recovery; spine surgery; intravenous lidocaine
MeSH Terms: conditions — Pain | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Active Comparator): Intravenous Lidocaine bolus of 1.5 mg/kg followed by infusion of 1.5 mg/kg/hr
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Normal saline placebo infusion
  Interventions: Other: Placebo (normal saline)

INTERVENTIONS:
Drug: Lidocaine — Lidocaine iv bolus followed by infusion
  Arms: Lidocaine
Other: Placebo (normal saline) — Normal saline bolus followed by infusion
  Arms: Placebo

SUMMARY:
Acute postoperative pain is an unpleasant, unwanted sensory and emotional experience for the patient. The investigators seek to determine if the addition of systemic lidocaine can improve the quality of recovery after spine surgery and reduce the requirement for opiate therapy.

DETAILED DESCRIPTION:
Consented patients will be randomized to either saline group or lidocaine group. General anesthesia will be induced as it would normally be done in any patient undergoing spine surgery. Once the patient is positioned for the surgery bolus followed by the infusion of either the study drug or the placebo will be administered. The infusion will be stopped at the end of surgery and the patient will be transferred to the post anesthesia care unit. Post operative pain score will be evaluated for the first 24 hrs and also the amount of pain medications used will be recorded. At the end of 24 hours quality of recovery will be assessed using a qor-40 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18-80 yrs;
2. American Society of Anesthesiology Physical Status I, II or III; and
3. Patients undergoing thoracic or lumbosacral spine surgeries with or without instrumentation via the posterior approach with planned admission to the post anesthesia care unit after surgery-

Exclusion Criteria:

1. Allergy to any of the study medications or anesthetic agents used in the study;
2. American Society of Anesthesiology physical status IV;
3. Spine surgery with the expected duration of surgery being more than 4 hours as determined by the attending surgeon;
4. History of severe hepatic dysfunction with liver enzymes elevated to more than 3 times the normal or International normalized ratio of more than 2 and renal dysfunction with GFR less than 60 ml/min
5. History of previous spinal fusion or instrumentation;
6. Diagnosis of cancer of the spine;
7. History of surgery for abscess or osteomyelitis;
8. History of cardiac dysrhythmia or heart block;
9. History of chronic heroin or methadone use;
10. Preoperative use of any systemic corticosteroid;
11. History of seizure disorder; and
12. Patient inability to properly describe postoperative pain to investigators (dementia, delirium, psychiatric disorder).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Quality of recovery | At 24 hours after surgery

SECONDARY OUTCOMES:
Post operative pain | for the first 24 hours after surgery

OTHER OUTCOMES:
Narcotic consumption | 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States